CLINICAL TRIAL: NCT07397260
Title: Effects of Manually Recorded or Automatically Transmitted Home Blood Pressures With or Without Automated Patient Feedback on Hypertension Care
Brief Title: Automatically Transmitted Home Blood Pressure and Automated Patient Feedback in Hypertension Care: the AUTO 2 Trial
Acronym: AUTO 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stephen Persell, MD, MPH, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STU00224615; R01HL179919 (NIH)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hypertension (HTN)
Keywords: Hypertension; Remote Patient Monitoring; RPM; Automated transmission; Home blood pressure; Hypertension Care
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Enhanced Usual Care (Active Comparator): Participants receive a blood pressure monitor and are encouraged to enter blood pressure results into their EHR patient portal.
  Interventions: Other: Self report of home measured blood pressure via patient EHR portal
- Automated Transmission of Remotely Monitored Blood Pressure (Active Comparator): Participants receive a blood pressure monitor and an application to directly transmit measurements to their EHR record.
  Interventions: Other: Automated Transmission of Remotely Measured Blood Pressure
- Automated Patient Feedback on Self Blood Pressure Monitoring (Active Comparator): Participants receive a blood pressure monitor and are encouraged to enter blood pressure results into their EHR patient portal. Participants receive messages through the EHR patient portal about their home blood pressure results.
  Interventions: Other: Self report of home measured blood pressure via patient EHR portal; Other: Automated feedback about home blood pressure results
- Automated Transmission of Remotely Monitored Blood Pressure and Automated Feedback (Active Comparator): Participants receive a blood pressure monitor and an application to directly transmit measurements to their EHR record. Participants receive messages through the EHR patient portal about their home blood pressure results.
  Interventions: Other: Automated feedback about home blood pressure results; Other: Automated Transmission of Remotely Measured Blood Pressure

INTERVENTIONS:
Other: Self report of home measured blood pressure via patient EHR portal — Participants will be provided with a home blood pressure monitor and method to use the EHR portal to enter home collected blood pressures into the EHR.
  Arms: Automated Patient Feedback on Self Blood Pressure Monitoring; Enhanced Usual Care
Other: Automated feedback about home blood pressure results — Patients will received periodic messages about the results of their home blood pressure monitoring with suggestions to consult with clinical care team when indicated.
  Arms: Automated Patient Feedback on Self Blood Pressure Monitoring; Automated Transmission of Remotely Monitored Blood Pressure and Automated Feedback
Other: Automated Transmission of Remotely Measured Blood Pressure — Participants will be provided with a blood pressure monitor and application to automatically transmit home blood pressures to their EHR record.
  Arms: Automated Transmission of Remotely Monitored Blood Pressure; Automated Transmission of Remotely Monitored Blood Pressure and Automated Feedback

SUMMARY:
The purpose of this study is to evaluate the effectiveness of automatically-generated medical advice to patients about to their home blood pressure monitoring results sent through patient portal messages compared to no automated advice and the effectiveness of automated transmission of remotely-obtained blood pressure values compared to self-reported values on systolic blood pressure at 1-year follow up in patients with uncontrolled hypertension whose physicians or advance practice providers provide primary care at Northwestern Medicine. Persistence of effects through 18 months will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-84 years at enrollment date
* Receives hypertension care primarily from a participating clinician
* Blood pressure on the two most recent days when ambulatory clinic blood pressure was obtained prior to patient identification to was ≥140 mm Hg systolic and/or ≥90 diastolic or last ambulatory clinic blood pressure was ≥150 mm Hg systolic and/or ≥95 diastolic
* Currently has or is willing to obtain a patient portal account from NM.

Exclusion Criteria:

* Dementia,
* Nursing home resident,
* Stage 5 chronic kidney disease or renal replacement therapy,
* Pregnancy,
* Receiving hospice,
* Not planning to continue to receive hypertension care from NM clinician for the next year,
* Planning to move from the region in the next year,
* Planning to change clinician treating their hypertension in the next year,
* Medical or psychological reason they cannot perform home blood pressure monitoring.
* Known to have average home blood pressure or most recent home blood pressure value of <130/80 mm Hg.

CLINICIAN PARTICIPANT INCLUSION Physician, advanced practice nurse or physician assistant working at a Northwestern Medicine ambulatory primary care site that cares for adults with hypertension (family medicine, internal medicine, medicine/pediatrics, and ambulatory geriatrics sites).

CLINICIAN PARTICIPANT EXCLUSION

* Primary care physicians and clinicians not willing for their patients to participate in study
* Planning to depart NM within the next year
* Not willing to receive patients' out-of-office blood pressure data

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1304 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure at 12 months | 12 months

SECONDARY OUTCOMES:
Systolic blood pressure at 18 months | 18 months
Antihypertensive medication changes from baseline | From baseline to 12 months and 18 months
Antihypertensive medication classes prescribed, standardized count | 12 months and 18 months
Medication adherence (patient report, Domains of Subjective Extent of Nonadhernece) | 12 months and 18 months
Diastolic blood pressure | 12 months and 18 months
Blood pressure <130/80 mm Hg | 12 months and 18 months
Blood pressure <140/90 mm Hg | 12 months and and 18 months

OTHER OUTCOMES:
Patient engagement (Consumer Health Activation Index) | 12 months and 18 months
Quality of Life (PROMIS® Scale v1.2 -Global Health) | 12 months and 18 months
Office encounters count | From baseline to 12 months and 18 months
Portal messages count | From baseline to 12 months and 18 months
Telephone encounters count at 1 year and 18 months | From baseline to 12 months and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Persell, MD,MPH, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Liu L, Shih YCT, Strawderman RL, Zhang DW, Johnson BA, Chai HT. Statistical Analysis of Zero-Inflated Nonnegative Continuous Data: A Review. Stat Sci. 2019;34(2):253-279
- [Background] HealthMeasures. PROMIS Scale v1.2 - Global Health. 2024. Available at https://www.healthmeasures.net/index.php?option=com_instruments&view=measure&id=778&Itemid=992.
- [Background] Condie RM, O'Reilly RJ. Prevention of cytomegalovirus infection in bone marrow transplant recipients by prophylaxis with an intravenous, hyperimmune cytomegalovirus globulin. Birth Defects Orig Artic Ser. 1984;20(1):327-44. No abstract available. PMID 6329370
- [Background] Voils CI, King HA, Thorpe CT, et al. Content Validity and Reliability of a Self-Report Measure of Medication Nonadherence in Hepatitis C Treatment. Dig Dis Sci. 2019;64(10):2784-2797
- [Background] Bartholomeusz RK, Bertoncello I. Anchorage-independence as an index of proliferative potential and maturational age: a comparison of the growth of normal, primary explanted bovine granulosa cells in semisolid agar and in liquid culture. Int J Cell Cloning. 1987 Mar;5(2):142-8. doi: 10.1002/stem.5530050206. PMID 3494794
- [Background] Cummings B. Empowering women: homoeopathy in midwifery practice. Complement Ther Nurs Midwifery. 1998 Feb;4(1):13-6. doi: 10.1016/s1353-6117(98)80007-3. PMID 9677928
- [Background] American Heart Association. Available at https://www.heart.org/en/health-topics/high-blood-pressure/understanding-blood-pressure-readings/monitoring-your-blood-pressure-at-home. 2024.
- [Background] Allen CE, Easley CE, Storfjell JI. Cost management through caseload/workload analysis. NLN Publ. 1986 Sep;(20-2155):331-46. No abstract available. PMID 3639439
- [Background] Il'ina TS. [A new type of potentially mobile genetic elements--integrons, assuring site-specific introduction of DNA modules with resistance genes, and expression of them]. Mol Gen Mikrobiol Virusol. 1993 Mar-Apr;(2):37-9. No abstract available. Russian. PMID 8390603
- [Background] Yamaguchi J, Kanematsu T, Shiku H, Nakayama E. Long-term survival of orthotopic Lewis liver grafts in Wistar Furth rats. Elimination or inactivation of effector CTL and altered antigenicity as possible reasons for tolerance. Transplantation. 1994 Feb;57(3):412-8. doi: 10.1097/00007890-199402150-00017. PMID 8108877
- [Background] Oliveria SA, Lapuerta P, McCarthy BD, L'Italien GJ, Berlowitz DR, Asch SM. Physician-related barriers to the effective management of uncontrolled hypertension. Arch Intern Med. 2002;162(4):413-420
- [Background] Weingarten JL, Cromie WJ, Paty RJ. Augmentation myoperitoneocystoplasty. J Urol. 1990 Jul;144(1):156-8. doi: 10.1016/s0022-5347(17)39400-4. PMID 2359169
- [Background] Rustia A, Wierzbicki V, Marrocco L, Tossini A, Zamponi C, Lista F. Is exon 5 of the PTEN/MMAC1 gene a prognostic marker in anaplastic glioma? Neurosurg Rev. 2001 Jul;24(2-3):97-102. doi: 10.1007/pl00014589. PMID 11485247
- [Background] Kerr EA, Zikmund-Fisher BJ, Klamerus ML, Subramanian U, Hogan MM, Hofer TP. The role of clinical uncertainty in treatment decisions for diabetic patients with uncontrolled blood pressure. Ann Intern Med. 2008;148(10):717-727
- [Background] Philipps KA Jr. Living wills--moral directive can cause legal dilemma. Hosp Med Staff. 1978 May;7(5):20-3. PMID 10236716
- [Background] Ehrenthal DB, Farber NJ, Collier VU, Aboff BM. Chaperone use by residents during pelvic, breast, testicular, and rectal exams. J Gen Intern Med. 2000 Aug;15(8):573-6. doi: 10.1046/j.1525-1497.2000.10006.x. PMID 10940150
- [Background] Kury G, Weiner J, Duval JV. Multiple self-inflicted gunshot wounds to the head: report of a case and review of the literature. Am J Forensic Med Pathol. 2000 Mar;21(1):32-5. doi: 10.1097/00000433-200003000-00005. PMID 10739223
- [Background] Pantoflickova D, Blum AL, Koelz HR. Helicobacter pylori and functional dyspepsia: a real causal link? Baillieres Clin Gastroenterol. 1998 Sep;12(3):503-32. doi: 10.1016/s0950-3528(98)90021-5. PMID 9890085
- [Background] Alarcon-Vargas D, Tansey WP, Ronai Z. Regulation of c-myc stability by selective stress conditions and by MEKK1 requires aa 127-189 of c-myc. Oncogene. 2002 Jun 27;21(28):4384-91. doi: 10.1038/sj.onc.1205543. PMID 12080469
- [Background] Becker H, Hartmann R, Kallmayer HJ, Lehr CM, Loth H, Maurer HH. [Pharmacy at the Univeristy of the Saarlands]. Pharm Unserer Zeit. 1997 Jul;26(4):199-201. doi: 10.1002/pauz.19970260408. No abstract available. German. PMID 9411452
- [Background] Persell SD. Reducing High-Risk Geriatric Polypharmacy Via EHR Nudges R01 Trial (HRPP), available at https://clinicaltrials.gov/study/NCT05656560?a=4.
- [Background] Rudduck GA, Harding GF. Visual electrophysiology to achromatic and chromatic stimuli in premature and full term infants. Int J Psychophysiol. 1994 May;16(2-3):209-18. doi: 10.1016/0167-8760(89)90048-2. PMID 8089040
- [Background] Gibson FS, Wei J, Vemishetti P, Gao Q, Dillon JL. Synthesis, utility, and X-ray crystal structure of novel complexes of baccatin III with imidazole and 2-propanol. Org Lett. 2000 Oct 19;2(21):3269-71. doi: 10.1021/ol006332q. PMID 11029187
- [Background] Persell SD, Brown T, Lee JY, et al. Individualized Risk Communication and Outreach for Primary Cardiovascular Disease Prevention in Community Health Centers: Randomized Trial. Circ Cardiovasc Qual Outcomes. 2015;8(6):560-566
- [Background] Clark CR, Davenport TW. Synthesis and anticonvulsant activity of analogues of 4-amino-N-(1-phenylethyl)benzamide. J Med Chem. 1987 Jul;30(7):1214-8. doi: 10.1021/jm00390a016. PMID 3599027
- [Background] Salzer H, Husslein P, Lohninger A, Binstorfer E, Langer M, Schonbauer M, Wagner G, Simbruner G, Popow C. [lst report: Alternatives to cortisone therapy. lst clinical experiences with a carnitine-betamethasone combination for the stimulation of fetal lung maturity]. Wien Klin Wochenschr. 1983 Oct 28;95(20):724-8. German. PMID 6689234
- [Background] Bendtzen K, Tvede N, Andersen V, Bendixen G. Cyclosporin for polymyositis. Lancet. 1984 Apr 7;1(8380):792-3. doi: 10.1016/s0140-6736(84)91301-1. No abstract available. PMID 6143105
- [Background] Zikrillaev Z, Gafarov ShS. [Calcified deferent duct simulating ureteral calculi]. Urologiia. 1999 Sep-Oct;(5):30-1. No abstract available. Russian. PMID 11150153
- [Background] Persell SD, Liss DT, Walunas TL, et al. Effects of 2 Forms of Practice Facilitation on Cardiovascular Prevention in Primary Care: A Practice-randomized, Comparative Effectiveness Trial. Med Care. 2020;58(4):344-351
- [Background] Azizi M, Sharp ASP, Fisher NDL, et al. Patient-Level Pooled Analysis of Endovascular Ultrasound Renal Denervation or a Sham Procedure 6 Months After Medication Escalation: The RADIANCE Clinical Trial Program. Circulation. 2024;149(10):747-759
- [Background] Bhatt DL, Kandzari DE, O'Neill WW, et al. A controlled trial of renal denervation for resistant hypertension. N Engl J Med. 2014;370(15):1393-1401
- [Background] Smith JM. Over-the-counter sale of antibiotics. N Z Med J. 1995 Jun 28;108(1002):258. No abstract available. PMID 7617336
- [Background] Schulz KF, Altman DG, Moher D, Group C. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010;152(11):726-732
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Background] Shah NJ, Unlu T, Wegener HP, Halling H, Zilles K, Appelt S. Measurement of rubidium and xenon absolute polarization at high temperatures as a means of improved production of hyperpolarized (129)Xe. NMR Biomed. 2000 Jun;13(4):214-9. doi: 10.1002/1099-1492(200006)13:43.0.co;2-g. PMID 10867699
- [Background] Borson DB, Chin RA, Davis B, Nadel JA. Adrenergic and cholinergic nerves mediate fluid secretion from tracheal glands of ferrets. J Appl Physiol Respir Environ Exerc Physiol. 1980 Dec;49(6):1027-31. doi: 10.1152/jappl.1980.49.6.1027. PMID 7440290
- [Background] Rotbart HA, Sawyer MH, Fast S, Lewinski C, Murphy N, Keyser EF, Spadoro J, Kao SY, Loeffelholz M. Diagnosis of enteroviral meningitis by using PCR with a colorimetric microwell detection assay. J Clin Microbiol. 1994 Oct;32(10):2590-2. doi: 10.1128/jcm.32.10.2590-2592.1994. PMID 7814507
- [Background] Acheson AL, Naujoks K, Thoenen H. Nerve growth factor-mediated enzyme induction in primary cultures of bovine adrenal chromaffin cells: specificity and level of regulation. J Neurosci. 1984 Jul;4(7):1771-80. doi: 10.1523/JNEUROSCI.04-07-01771.1984. PMID 6145760
- [Background] Trkulja V, Lackovic Z. [Ecstasy]. Lijec Vjesn. 1997 May-Jun;119(5-6):158-66. Croatian. PMID 9379824
- [Background] Murdoch ME, Payton A, Abiose A, Thomson W, Panicker VK, Dyer PA, Jones BR, Maizels RM, Ollier WE. HLA-DQ alleles associate with cutaneous features of onchocerciasis. The Kaduna-London-Manchester Collaboration for Research on Onchocerciasis. Hum Immunol. 1997 Jun;55(1):46-52. doi: 10.1016/s0198-8859(97)00089-x. PMID 9328789
- [Background] Chalom S, Elrezzi E, Pena P, Astiarsaran I, Bello J. Composition of sulfited potatoes: comparison with fresh and frozen potatoes. Plant Foods Hum Nutr. 1995 Feb;47(2):133-8. doi: 10.1007/BF01089262. PMID 7792261
- [Background] Fowler SB, Cicoca R, Keller I. Patient care following carotid endarterectomy. Medsurg Nurs. 1999 Feb;8(1):47-52. PMID 10232212
- [Background] Centers for Medicare and Medicaid Services Federal Register/Vol. 84, No. 221/Friday, November 15, 2019/Rules and Regulations. 42 CFR Parts 403, 409, 410, 411, 414, 415, 416, 418, 424, 425, 489, and 498 [CMS-1715-F and IFC].
- [Background] Lin M, Napoli JL. cDNA cloning and expression of a human aldehyde dehydrogenase (ALDH) active with 9-cis-retinal and identification of a rat ortholog, ALDH12. J Biol Chem. 2000 Dec 22;275(51):40106-12. doi: 10.1074/jbc.M008027200. PMID 11007799
- [Background] Lopez-Bote CJ, Gray JI, Gomaa EA, Flegal CJ. Effect of dietary administration of oil extracts from rosemary and sage on lipid oxidation in broiler meat. Br Poult Sci. 1998 May;39(2):235-40. doi: 10.1080/00071669889187. PMID 9649877
- [Background] Sultan PG, Ganley TJ, Carpentieri DF, Harty MP. Draining sinus of the upper arm in a 12-year-old girl. Clin Orthop Relat Res. 2000 Sep;(378):312-6, 319-22. doi: 10.1097/00003086-200009000-00042. No abstract available. PMID 10987007
- [Background] Ch'ien LT, Halsey JH Jr. Trigeminal sensory neuropathy and bell's palsy. N Engl J Med. 1970 Jan 22;282(4):224-5. doi: 10.1056/NEJM197001222820414. No abstract available. PMID 4311883
- [Background] Dittmer A. [Use of antibiotics--principles and possibilities]. Z Gesamte Hyg. 1984 Jan;30(1):2-7. No abstract available. German. PMID 6324502
- [Background] Mills A. Economic evaluation of health programmes: application of the principles in developing countries. World Health Stat Q. 1985;38(4):368-82. No abstract available. English, French. PMID 3938109
- [Background] Magid DJ, Olson KL, Billups SJ, Wagner NM, Lyons EE, Kroner BA. A pharmacist-led, American Heart Association Heart360 Web-enabled home blood pressure monitoring program. Circ Cardiovasc Qual Outcomes. 2013;6(2):157-163
- [Background] Yamaguchi H, Iwata K. [Dimorphism and cell wall structure of fungi]. Tanpakushitsu Kakusan Koso. 1972 Aug;17(8):588-603. No abstract available. Japanese. PMID 4565195
- [Background] Bosworth HB, Powers BJ, Olsen MK, et al. Home blood pressure management and improved blood pressure control: results from a randomized controlled trial. Arch Intern Med. 2011;171(13):1173-1180
- [Background] Pierau H. [Solid waste materials]. Offentl Gesundheitswes. 1972 Dec;34:Suppl 2:73-6. No abstract available. German. PMID 4266385
- [Background] Ma L, Pu MY, Yi H, Akhand AA, Ohata N, Ohkusu K, Kato M, Iwamoto T, Isobe K, Hamaguchi M, et al. Multiphasic modulation of signal transduction into T lymphocytes by monoiodoacetic acid as a sulfhydryl reagent. J Cell Biochem. 1995 Sep;59(1):33-41. doi: 10.1002/jcb.240590105. PMID 8530534
- [Background] McManus RJ, Mant J, Haque MS, et al. Effect of self-monitoring and medication self-titration on systolic blood pressure in hypertensive patients at high risk of cardiovascular disease: the TASMIN-SR randomized clinical trial. JAMA. 2014;312(8):799-808
- [Background] McManus RJ, Mant J, Bray EP, et al. Telemonitoring and self-management in the control of hypertension (TASMINH2): a randomised controlled trial. Lancet. 2010;376(9736):163-172
- [Background] Horio T, Kawamura Y. Effects of texture of food on chewing patterns in the human subject. J Oral Rehabil. 1989 Mar;16(2):177-83. doi: 10.1111/j.1365-2842.1989.tb01331.x. PMID 2715866
- [Background] Wakefield BJ, Holman JE, Ray A, et al. Effectiveness of home telehealth in comorbid diabetes and hypertension: a randomized, controlled trial. Telemed J E Health. 2011;17(4):254-261
- [Background] Burdine JA Jr, Werch A. 113mIn gelatin complex for placental localization. Am J Obstet Gynecol. 1969 Jul 1;104(5):748-51. doi: 10.1016/0002-9378(69)90620-6. No abstract available. PMID 5788021
- [Background] Volynskii ZM. [The current status of knowledge in the field of arteriosclerosis]. Voen Med Zh. 1967 Jan;1:14-9. No abstract available. Russian. PMID 5604965
- [Background] Morrison R, Shovlin JP. A review of the use of bandage lenses. Metab Pediatr Syst Ophthalmol. 1982;6(2):117-21. No abstract available. PMID 7162426
- [Background] Bugaenko NN, Gorban' AN, Sadovskii MG. [Determination of the amount of information in nucleotide sequences]. Mol Biol (Mosk). 1996 May-Jun;30(3):529-41. No abstract available. Russian. PMID 8754001
- [Background] Stergiou GS, Kollias A, Zeniodi M, Karpettas N, Ntineri A. Home blood pressure monitoring: primary role in hypertension management. Curr Hypertens Rep. 2014;16(8):462
- [Background] Lu Y, Linderman GC, Mahajan S, et al. Quantifying Blood Pressure Visit-to-Visit Variability in the Real-World Setting: A Retrospective Cohort Study. Circ Cardiovasc Qual Outcomes. 2023;16(4):e009258
- [Background] Campbell NR, Culleton BW, McKay DW. Misclassification of blood pressure by usual measurement in ambulatory physician practices. Am J Hypertens. 2005;18(12 Pt 1):1522-1527
- [Background] Stergiou GS. How to cope with unreliable office blood pressure measurement? Am J Hypertens. 2005;18(12 Pt 1):1519-1521
- [Background] Watanabe T, Honda Y, Fujii Y, Koyama M, Matsuzawa H, Tanaka R. Three-dimensional anisotropy contrast magnetic resonance axonography to predict the prognosis for motor function in patients suffering from stroke. J Neurosurg. 2001 Jun;94(6):955-60. doi: 10.3171/jns.2001.94.6.0955. PMID 11409525
- [Background] Bovre K. Oxidase positive bacteria in the human nose incidence and species distribution, as diagnosed by genetic transformation. Acta Pathol Microbiol Scand B Microbiol Immunol. 1970;78(6):780-4. No abstract available. PMID 5278896
- [Background] Whelton PK, Carey RM, Aronow WS, et al. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2018;71(19):e127-e248
- [Background] Panagiotakos D, Antza C, Kotsis V. Ambulatory and home blood pressure monitoring for cardiovascular disease risk evaluation: a systematic review and meta-analysis of prospective cohort studies. J Hypertens. 2024;42(1):1-9
- [Background] Kollias A, Kyriakoulis KG, Komnianou A, Stathopoulou P, Stergiou GS. Prognostic value of home versus ambulatory blood pressure monitoring: a systematic review and meta-analysis of outcome studies. J Hypertens. 2024;42(3):385-392
- [Background] Krist AH, Davidson KW, et al. Screening for Hypertension in Adults: US Preventive Services Task Force Reaffirmation Recommendation Statement. JAMA. 2021;325(16):1650-1656
- [Background] Loewenstein-Lichtenstein Y, Schwarz M, Glick D, Norgaard-Pedersen B, Zakut H, Soreq H. Genetic predisposition to adverse consequences of anti-cholinesterases in 'atypical' BCHE carriers. Nat Med. 1995 Oct;1(10):1082-5. doi: 10.1038/nm1095-1082. PMID 7489367
- [Background] Aguilar MI, Saez J, Llorens M, Soler A, Ortuno JF. Nutrient removal and sludge production in the coagulation-flocculation process. Water Res. 2002 Jun;36(11):2910-9. doi: 10.1016/s0043-1354(01)00508-5. PMID 12146881